CLINICAL TRIAL: NCT00919204
Title: An Open Label Phase 1 Study To Evaluate The Pharmacokinetics Of AG-013736 In Healthy Chinese Volunteers
Brief Title: Axitinib Pharmacokinetics in Chinese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: A4061050
Record Dates: First submitted 2009-06-11; First posted 2009-06-12 (Estimated); Last update posted 2009-09-21 (Estimated); Status verified 2009-09

CONDITIONS: Healthy Volunteers
Keywords: AG-013736, axitinib, pharmacokinetics, healthy, Chinese
MeSH Terms: interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort 1 (Experimental)
  Interventions: Drug: AG-013736 (axitinib)

INTERVENTIONS:
Drug: AG-013736 (axitinib) — Three single oral-doses of AG-013736 (5-mg, 7-mg and 10-mg) will be successively administered (each separated by a washout period of at least 7 days) to healthy Chinese volunteers in the fed state.

SUMMARY:
As part of the global clinical development program for AG-013736, studies are ongoing (and planned) in cancer patients in China. An assessment of AG-013736 pharmacokinetics in Chinese subjects, as required by the Chinese Health Authorities, is therefore warranted.

In the current study the single dose pharmacokinetics of AG-013736 will be characterized at 3 doses (5 mg, 7 mg and 10 mg).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female (of nonchildbearing potential) Chinese (individuals currently residing in mainland China who were born in China and have both parents of Chinese descent) subjects between the ages of 18 and 45 years, inclusive. (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests.)
* Body Mass Index (BMI) of 19 to 24 kg/m2; and a total body weight >50 kg (110 lbs). A BMI lower limit of 18.5 kg/m2 may be rounded up to 19.0 kg/m2; a BMI upper limit of 24.5 kg/m2 may be rounded down to 24.0 kg/m2 and will be acceptable for inclusion.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) disease or clinical findings at Screening.
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* Drug dependency, a positive urine drug screen, or alcohol dependency.
* History of regular alcohol consumption exceeding 28 or more units per week. (One unit=285 mL of beer or 25 mL of spirits or 125 mL of wine).
* Use of tobacco- or nicotine-containing products (or a positive urine cotinine test).
* Treatment with an investigational drug within 3 months (or as determined by local regulations) or 5 half-lives preceding the first dose of study medication.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2009-08; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Plasma Pharmacokinetics of AG-013736 in Chinese Healthy Volunteers | 3 months

SECONDARY OUTCOMES:
Safety of AG-013736 in Chinese Healthy Volunteers | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Beijng, China

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4061050&StudyName=Axitinib%20Pharmacokinetics%20in%20Chinese%20Healthy%20Volunteers